CLINICAL TRIAL: NCT07233616
Title: Risks and Benefits of Radiofrequency Ablation for Chronic Venous Insufficiency (CEAP C3-C6) in Patients Aged 80 and Over: A Prospective Single-Arm Cohort Study
Brief Title: Risks and Benefits of Radiofrequency Ablation for Chronic Venous Insufficiency (CEAP C3-C6) in Patients Aged 80 and Over
Status: Recruiting | Type: Observational
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunshui He, chief physician, Chengdu University of Traditional Chinese Medicine
Other Study IDs: ChengduUTCM 121
Record Dates: First submitted 2025-09-28; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Chronic Venous Insufficiency, CVI; Radiofrequency Ablation; Octogenarians(Aged 80 and Over); Cohort Study
MeSH Terms: conditions — Blindness, Cortical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endovenous Radiofrequency Ablation — All patients undergo endovenous radiofrequency ablation(RFA) under local tumescent anesthesia. Using the ClosureFast™ system (or equivalent), the target saphenous vein is accessed percutaneously under ultrasound guidance. After catheter placement and tumescent anesthesia infiltration, radiofrequency energy is delivered segmentally to ablate the vein. Post-procedure, compression bandaging is applied and Class II compression stockings are prescribed.

SUMMARY:
The prevalence of severe chronic venous insufficiency (CVI) is significant in the growing octogenarian population. While radiofrequency ablation (RFA) is a standard minimally invasive treatment, robust data on its outcomes and safety profiles specifically in patients aged 80 years and older remain scarce. This study aims to evaluate the risks and benefits of RFA in this specific, high-risk demographic.This prospective, single-arm, single-center cohort study will enroll 50 patients (initial target sample size) aged ≥80 years with CVI classified as CEAP C3 to C6 and with confirmed great or small saphenous vein reflux. All participants will undergo endovenous RFA under tumescent local anesthesia. The primary outcomes are: 1) the great/small saphenous vein occlusion rate at 6 months, assessed by duplex ultrasonography, and 2) the change in disease-specific quality of life from baseline to 6 months, measured by the Aberdeen Varicose Vein Questionnaire (AVVQ). Secondary outcomes include occlusion rates at 1 and 3 months; complication rates (e.g., deep vein thrombosis, skin burns, paresthesia) within 30 days; and changes in the Venous Clinical Severity Score (VCSS) and the 12-Item Short Form Health Survey (SF-12) at predefined intervals over 6 months.This study is designed to demonstrate a high technical success rate (occlusion rate >95% at 6 months) and a statistically significant improvement in AVVQ and VCSS scores at 6 months post-procedure. The collected data will provide a detailed profile of complication rates, characterizing the safety of RFA in this very elderly cohort.This study will provide crucial, prospective evidence regarding the efficacy and safety of RFA for treating CVI in octogenarians. The findings are expected to guide clinical decision-making and inform treatment guidelines for this vulnerable and expanding patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Aged 80 years or older.
2. Clinical Diagnosis: Symptomatic chronic venous insufficiency of the lower extremity, with the highest clinical class (CEAP classification) being one of the following:

   * C3: Venous edema
   * C4a: Pigmentation or eczema
   * C4b: Lipodermatosclerosis or atrophie blanche
   * C5: Healed venous ulcer
   * C6: Active venous ulcer
3. Confirmed Reflux: Color duplex ultrasound examination confirming reflux (reflux time > 0.5 seconds) in the great saphenous vein (GSV) and/or small saphenous vein (SSV) of the target limb.
4. Informed Consent: The patient or their legally authorized representative is able to understand and voluntarily provides written informed consent.

Exclusion Criteria:

* Participants who meet any of the following criteria will be excluded from the study:

  1. Mobility: Non-ambulatory or bedridden.
  2. Thrombosis: Presence of acute superficial thrombophlebitis of the target vein, or deep vein thrombosis (DVT) in the target limb.
  3. Arterial Disease: Significant peripheral arterial disease, defined as an ankle-brachial index (ABI) < 0.8 in the target limb.
  4. Coagulopathy: Uncorrectable coagulation disorder.
  5. Allergy: Known severe allergy to local anesthetics (e.g., lidocaine) or relevant device materials.
  6. Cognition & Compliance: Severe cognitive impairment or psychiatric illness that, in the investigator's judgment, precludes adequate understanding and cooperation for the study procedures and follow-up.
  7. Life Expectancy: Life expectancy of less than 1 year due to other comorbid conditions (e.g., terminal malignancy).
  8. General Unsuitability: Any other condition that, in the opinion of the investigator, makes the patient unsuitable for participation in the study.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consists of patients aged 80 years and older who are diagnosed with symptomatic, severe chronic venous insufficiency (CVI), classified as CEAP clinical classes C3 through C6, and have confirmed great or small saphenous vein reflux.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Great/Small Saphenous Vein Occlusion Rate at 6 Months | 6 Months
Aberdeen Varicose Vein Questionnaire (AVVQ) | 6 Months
  Minimum Score: 0 Maximum Score: 100 Interpretation of Higher Scores: A higher score indicates more severe symptom distress and greater impact on quality of life caused by varicose veins in patients. For example, it reflects more obvious discomforts such as leg pain, a heavy sensation in the legs, and swelling.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kulkarni SR, Slim FJ, Emerson LG, Davies C, Bulbulia RA, Whyman MR, Poskitt KR. Effect of foam sclerotherapy on healing and long-term recurrence in chronic venous leg ulcers. Phlebology. 2013 Apr;28(3):140-6. doi: 10.1258/phleb.2011.011118. PMID 22422794
- [Result] Williamsson C, Danielsson P, Smith L. Catheter-directed foam sclerotherapy for chronic venous leg ulcers. Phlebology. 2014 Dec;29(10):688-93. doi: 10.1177/0268355513505506. Epub 2013 Sep 26. PMID 24072751
- [Result] Mohamed AH, Howitt A, Rae S, Cai PL, Hitchman L, Wallace T, Nandhra S, Pymer S, Knighton A, Smith G, Chetter IC, Carradice D. Ten-year outcomes of a randomized clinical trial of endothermal ablation versus conventional surgery for great saphenous varicose veins. Br J Surg. 2024 Aug 2;111(8):znae195. doi: 10.1093/bjs/znae195. PMID 39162334